CLINICAL TRIAL: NCT06705491
Title: Trauma-Informed Procedural Pain Intervention: Refinement of an Evidence-Based Protocol
Acronym: TIPPI-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Kentucky Cabinet for Health and Family Services (Unknown); University of Kentucky (Other); Norton Healthcare (Other)
Responsible Party: Principal Investigator, Lauren Hayes, Assistant Professor, Department of Pediatrics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24.0284
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Procedural Pain; Cancer-related Pain
MeSH Terms: conditions — Pain, Procedural; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TIPPI-R (Experimental)
  Interventions: Behavioral: TIPPI-R
- Standard of Care (No Intervention): Participants and families in this arm will receive the standard treatment for pain and distress during cancer treatment at each respective institution, which may include psychoeducation and support implementing pain coping skills from mental health providers within the healthcare system.
- Delayed Intervention Delivery (Experimental): Participants will be moved into this arm if they are initially randomized into the intervention arm, but they receive the TIPPI-R intervention outside of the window dictated in the protocol. According to the protocol, consented participants should receive the interventions within 2 weeks of consent. If they do not, the TIPPI-R intervention will still be delivered and the participant will be moved to this arm of the study.
  Interventions: Behavioral: TIPPI-R

INTERVENTIONS:
Behavioral: TIPPI-R — The TIPPI-R intervention protocol consists of a one session, during which time the interventionist offers psychoeducation related to the following content areas: procedural pain related to oncology treatment, factors that may affect the perception of pain, evidenced-based tools for assessing and monitoring pain, cognitive and behavioral pain management interventions, and resources to facilitate family to advocacy for pain management in a medical setting. During this session, the interventionist discusses opportunities for families to utilize skills throughout treatment, and addresses family questions as needed. A follow-up session 4 weeks after the initial intervention session will assess family knowledge and skills and offer a referral for a mental health provider, if further pain management support is needed. TIPPI-R is designed to be delivered by a psychologist, psychology trainee, or social worker working in the oncology context.
  Arms: Delayed Intervention Delivery; TIPPI-R

SUMMARY:
The Trauma-Informed Procedural Pain Intervention (TIPPI-R) has been developed as a standardized way to provide education and teach evidence-based strategies for managing pain and distress that may occur during pediatric cancer treatment. The purpose of this clinical trial study is to test how helpful TIPPI-R is in supporting children and families manage pain and distress during the initial stages of cancer treatment. The main questions this study aims to answer are:

* Does TIPPI-R increase use of helpful pain coping strategies for pediatric cancer patients?
* Does TIPPI-R help lower perceived pain intensity during initial stages of cancer treatment?
* Does TIPPI-R increase patient and family confidence in coping with pain and distress during cancer treatment?

Researchers will compare pain experiences and use of pain coping strategies for families who receive the TIPPI-R intervention and families who receive standard of care to see if TIPPI-R decrease pain and distress during the initial stages of cancer treatment.

Participants will:

* Complete surveys to measure pain and distress within 5 weeks of initial diagnosis (Time 1)
* Either receive the TIPPI-R intervention or standard of care
* Complete surveys to measure pain and distress 4 weeks after initial consent or TIPPI-R intervention delivery (Time 2)

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving treatment at Norton Children's Cancer Institute, Norton Children's Hospital, University of Kentucky Children's Hospital or DanceBlue Clinic.
* Patient has been diagnosed with an oncology diagnosis.
* Patient and family are English-speaking.
* Patient is between the ages 0-18.

Exclusion Criteria:

* Families not proficient in English.
* Patient is 19 years or older.
* Patient is not receiving treatment at Norton Children's Cancer Institute, Norton Children's Hospital, University of Kentucky Children's Hospital or DanceBlue Clinic.
* Patient does not have an oncology diagnosis.
* Patient and family have any CPS involvement.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Coping Strategies | Pain coping strategies will be assessed at baseline (Time 1) and again approximately 4-6 weeks after being consented (Time 2).
  Families who receive TIPPI-R will report greater use of adaptive pain coping strategies than families in the standard of care condition. This is measured by Survey of Pain Management Practices, Pain Coping Questionnaire-Short Form (Parent and Child), and data abstraction from medical charts. The Survey of Pain Management Practices indicates how often pain management strategies are used over the past 7 days (or since diagnosis). Frequencies are rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Scores are calculated by summing the number of strategies used, with higher scores indicating greater frequency of use of adaptive coping strategies. The Pain Coping Questionnaire-Short Form (Child and Parent version) is a 16-item measure to assess how children cope with pain. Items are ranked on a 5-point Likert scale ranging from 1 (never) to 5 (very often). A mean scale score is calculated for each subscale, with higher scores indicating more of the measured construct.

SECONDARY OUTCOMES:
Perceived Pain Intensity | Perceived pain intensity will be assessed at baseline (Time 1) and again approximately 4-6 weeks after being consented (Time 2).
  Patients and families who receive TIPPI-R will report lower perceived intensity of pain experienced by patient than patients and families in the standard of care condition. This outcome will be measured by the Child Pain Characteristics Survey. Children and parent proxy rate worst, least, and average pain over the last 7 days on a scale from 0 (no pain) to 10 (worst possible pain), identify the location(s) of the pain, and indicate what they believe to be the source(s) of the pain.
Pain Catastrophizing | Pain catastrophizing will be assessed at baseline (Time 1) and again approximately 4-6 weeks after being consented (Time 2).
  Patients and families who receive TIPPI-R will report lower rates of pain catastrophizing than patients and families in the standard of care condition. This outcome will be measured by the Pain Catastrophizing Questionnaire-Parent and Child forms. These forms each include13 items across 3 subscales (rumination, magnification, and helplessness), which assess children's catastrophic thoughts and feelings about their pain. Raters indicate the extent to which they/their child experience each of the items using a 5-point Likert type scale ranging from not at all to extremely, with a higher score indicating more catastrophic thinking.
Confidence Managing Pain and Distress | Confidence managing pain and distress will be assessed at baseline and again approximately 4-6 weeks after being consented (Time 2).
  Patients and families who receive TIPPI-R will report higher confidence facilitating patient coping with pain and distress than families in the treatment as usual condition. This outcome will be measured by the Confidence in Pain Management measure. The child/caregiver will rate three questions on a scale from 0 (not at all confident) to 10 (very confident). Higher numerical rating will indicate greater confidence in pain management.
Distress | Distress will be assessed at baseline and again approximately 4-6 weeks after being consented (Time 2).
  Patients and families who receive TIPPI-R will report lower levels of distress than families in the treatment as usual condition. This outcome will be measured by the Emory Distress Thermometer. Caregiver and child (8 years and older) distress will be measured with 1 item, in which caregivers and patients will each indicate the degree of distress they have been experiencing in the past week ranging from 0 (no distress) to 10 (extreme distress).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren R Hayes, PhD, Principal Investigator — Norton Children's Medical Group, Affiliated with the University of Louisville School of Medicine
Locations (4):
- United States (4):
  - UK DanceBlue Pediatric Hematology & Oncology, Lexington, Kentucky
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Cancer Institute, Louisville, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tutelman PR, Chambers CT, Stinson JN, Parker JA, Fernandez CV, Witteman HO, Nathan PC, Barwick M, Campbell F, Jibb LA, Irwin K. Pain in Children With Cancer: Prevalence, Characteristics, and Parent Management. Clin J Pain. 2018 Mar;34(3):198-206. doi: 10.1097/AJP.0000000000000531. PMID 28678061
- [Background] O'Donnell FT, Rosen KR. Pediatric pain management: a review. Mo Med. 2014 May-Jun;111(3):231-7. PMID 25011346
- [Background] Tonning Olsson I, Alberts NM, Li C, Ehrhardt MJ, Mulrooney DA, Liu W, Pappo AS, Bishop MW, Anghelescu DL, Srivastava D, Robison LL, Hudson MM, Ness KK, Krull KR, Brinkman TM. Pain and functional outcomes in adult survivors of childhood cancer: A report from the St. Jude Lifetime Cohort study. Cancer. 2021 May 15;127(10):1679-1689. doi: 10.1002/cncr.33303. Epub 2020 Dec 28. PMID 33369896
- [Background] Schwartz LA, Brumley LD. What a Pain: The Impact of Physical Symptoms and Health Management on Pursuit of Personal Goals Among Adolescents with Cancer. J Adolesc Young Adult Oncol. 2017 Mar;6(1):142-149. doi: 10.1089/jayao.2016.0031. Epub 2016 Oct 28. PMID 27792462
- [Background] Price J, Kassam-Adams N, Alderfer MA, Christofferson J, Kazak AE. Systematic Review: A Reevaluation and Update of the Integrative (Trajectory) Model of Pediatric Medical Traumatic Stress. J Pediatr Psychol. 2016 Jan-Feb;41(1):86-97. doi: 10.1093/jpepsy/jsv074. Epub 2015 Aug 28. PMID 26319585
- [Background] Rosenberg AR, Bradford MC, Junkins CC, Taylor M, Zhou C, Sherr N, Kross E, Curtis JR, Yi-Frazier JP. Effect of the Promoting Resilience in Stress Management Intervention for Parents of Children With Cancer (PRISM-P): A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911578. doi: 10.1001/jamanetworkopen.2019.11578. PMID 31532518
- [Background] Kearney JA, Salley CG, Muriel AC. Standards of Psychosocial Care for Parents of Children With Cancer. Pediatr Blood Cancer. 2015 Dec;62 Suppl 5(Suppl 5):S632-83. doi: 10.1002/pbc.25761. PMID 26700921
- [Background] Uhl K, Burns M, Hale A, Coakley R. The Critical Role of Parents in Pediatric Cancer-Related Pain Management: a Review and Call to Action. Curr Oncol Rep. 2020 Mar 14;22(4):37. doi: 10.1007/s11912-020-0899-7. PMID 32172378
- [Background] Marsac ML, Kassam-Adams N, Hildenbrand AK, Nicholls E, Winston FK, Leff SS, Fein J. Implementing a Trauma-Informed Approach in Pediatric Health Care Networks. JAMA Pediatr. 2016 Jan;170(1):70-7. doi: 10.1001/jamapediatrics.2015.2206. PMID 26571032
- [Background] Stehl ML, Kazak AE, Alderfer MA, Rodriguez A, Hwang WT, Pai AL, Boeving A, Reilly A. Conducting a randomized clinical trial of an psychological intervention for parents/caregivers of children with cancer shortly after diagnosis. J Pediatr Psychol. 2009 Sep;34(8):803-16. doi: 10.1093/jpepsy/jsn130. Epub 2008 Dec 17. PMID 19091806
- [Background] Kazak AE, Hocking MC, Ittenbach RF, Meadows AT, Hobbie W, DeRosa BW, Leahey A, Kersun L, Reilly A. A revision of the intensity of treatment rating scale: classifying the intensity of pediatric cancer treatment. Pediatr Blood Cancer. 2012 Jul 15;59(1):96-9. doi: 10.1002/pbc.23320. Epub 2011 Aug 19. PMID 21858914
- [Background] Stinson JN, Jibb LA, Nguyen C, Nathan PC, Maloney AM, Dupuis LL, Gerstle JT, Hopyan S, Alman BA, Strahlendorf C, Portwine C, Johnston DL. Construct validity and reliability of a real-time multidimensional smartphone app to assess pain in children and adolescents with cancer. Pain. 2015 Dec;156(12):2607-2615. doi: 10.1097/j.pain.0000000000000385. PMID 26580680
- [Background] Kohut SA, Stinson J, Chambers CT, Reid GJ, Pillai Riddell RR. The Pain Coping Questionnaire short-form: preliminary reliability and validity. Pain Rep. 2022 Jan 12;7(1):e982. doi: 10.1097/PR9.0000000000000982. eCollection 2022 Jan-Feb. PMID 35047713
- [Background] Reid GJ, Gilbert CA, McGrath PJ. The Pain Coping Questionnaire: preliminary validation. Pain. 1998 May;76(1-2):83-96. doi: 10.1016/s0304-3959(98)00029-3. PMID 9696461
- [Background] Goubert L, Eccleston C, Vervoort T, Jordan A, Crombez G. Parental catastrophizing about their child's pain. The parent version of the Pain Catastrophizing Scale (PCS-P): a preliminary validation. Pain. 2006 Aug;123(3):254-263. doi: 10.1016/j.pain.2006.02.035. Epub 2006 Apr 27. PMID 16644128
- [Background] Caes L, Goubert L, Devos P, Verlooy J, Benoit Y, Vervoort T. The relationship between parental catastrophizing about child pain and distress in response to medical procedures in the context of childhood cancer treatment: a longitudinal analysis. J Pediatr Psychol. 2014 Aug;39(7):677-86. doi: 10.1093/jpepsy/jsu034. Epub 2014 Jun 6. PMID 24906963
- See also: Key Ingredients for Successful Trauma-Informed Care Implementation — https://www.samhsa.gov/sites/default/files/programs_campaigns/childrens_mental_health/atc-whitepaper-040616.pdf